CLINICAL TRIAL: NCT06448494
Title: Evaluation of the New Peri-Operative Geriatric Units in Ile-de-France, in Digestive and Urological Surgery
Acronym: UPOG-DIGU
Status: Recruiting | Type: Observational
Sponsor: Gérond'if (Other)
Responsible Party: Sponsor
Other Study IDs: 2022-A02302-41
Record Dates: First submitted 2024-06-04; First posted 2024-06-07 (Actual); Last update posted 2024-06-07 (Actual); Status verified 2024-06

CONDITIONS: Digestive and Urological Surgery
Keywords: Digestive and Urological Surgery; Peri-operative geriatric unit

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Prospective group: Patients who recieved geriatric perioperative car
- Retrospective group: Patients who received standard surgical care

SUMMARY:
The main objective of this study is to evaluate the effectiveness of experimental management by digestive or urological "new Peri-Operative Geriatric Units", on post-operative follow-up in the 3 months following the procedure.

Medical follow-up in the 10 days following the operation up to discharge, and patient outcomes in the 3 months following the operation, will be documented.

These data will be compared with data from subjects operated on in the reference year.

DETAILED DESCRIPTION:
This is a multicenter, non-interventional, prospective retrospective study:

* Prospective group: inclusion of patients scheduled to undergo one of the 9 procedures targeted by the "new Peri-Operative Geriatric Units" trial (colectomy, cholecystectomy, , transurethral prostatectomy, transurethral or transcutaneous procedure for non-lithiasis conditions, kidney and ureter procedure and major bladder surgery for tumor condition esophageal, gastric and duodenal procedure for malignancy, transurethral bladder resection)
* Retrospective group: inclusion of patients who were operated in 2019

This study will assess whether "Peri-Operative Geriatric Units" for digestive or urinary surgery is beneficial for :

* Medical follow-up in the 10 days following the operation and up to discharge (simple follow-up, complications, return to the operating room, etc.),
* Patient outcomes in the 3 months following surgery (discharge date, geriatric assessment, rehospitalization, other significant medical events, etc.).

These data will be compared with those of patients operated on in the reference year prior to pandemic Covid-19 (2019), who unlike you will not have benefited from "new Peri-Operative Geriatric Units" care.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subject, aged ≥ 75 years,
* Subject receiving or having received one of the 9 procedures targeted by the study: colectomy, or cholecystectomy, or nephrectomy, or transurethral resection of prostate adenoma, or transurethral prostatectomy, or transurethral or transcutaneous surgery for non-lithiasis conditions, or kidney and ureter surgery and major bladder surgery for tumor disease, or esophageal, stomach and duodenal surgery for malignancy, or transurethral resection of bladder,
* Subject orally agreeing (non-opposition), after having been informed and having been given a reasonable period of reflection, to participate in the study.

Exclusion Criteria:

* Patient having to undergo, at the time the study is proposed and over the theoretical period of participation, one or more other interventions already scheduled (other than the 9 mentioned in the inclusion criteria), and which, in the investigator's opinion, could have an impact on the study indicators7
* Subject unable to understand the purpose of the research, to answer questions and to give his/her decision to participate in the study,
* Subjects under legal protection or unable to express their consent, in accordance with article L1121-8 of the French Public Health Code,
* Subject already included in another research project involving the human body,
* Subject not affiliated to or not benefiting from a social security scheme.

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Elderly patients scheduled to undergo one of the 4 procedures targeted by the study (colectomy, or cholecystectomy, or nephrectomy, or transurethral resection of prostate adenoma)
Sampling Method: Non-Probability Sample
Enrollment: 1400 (Estimated)
Dates: Start 2023-05-31 (Actual); Primary Completion 2025-02-28 (Estimated); Study Completion 2025-08-28 (Estimated)

PRIMARY OUTCOMES:
Assessment of the effectiveness of experimental management by geriatric peri-operative digestive or urological units | 3 months

SECONDARY OUTCOMES:
Assessment of commorbidity risk according Charlson Comorbidity Index (CCI) | At inclusion
  The Charlson Comorbidity Index (CCI) assesses the level of comorbidity by considering the level of severity of 19 predefined comorbid disorders and the number of disorders present among them.
Assessment of the degree of patient dependence according Katz Index of Independence in Activities of Daily Living (ADL) | 3 months
  Katz Index of Independence in Activities of Daily Living is an unabbreviated scale title.
  This Index ranks adequacy of performance in the six functions of bathing, dressing, toileting, transferring, continence, and feeding. Patients are scored yes/no for independence in each of the six functions. A score of 6 indicates full function, 4 indicates moderate impairment, and 2 or less indicates severe functional impairment.
Assessment of patient's level of dependence through an appreciation of instrumental activities of daily living according Lawton scale | 3 months
Screening for a nutritional disorder according Body Mass Index (BMI) score | 3 months
Assessment of a patient's pre-operative state of health according The American Society of Anaesthesiologists score (ASA) | 3 months
  To determine if patient is healthy enough to tolerate surgery and anesthesia

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Hanon, PhD, MPH, Study Chair — Geriatric Departement, Broca Hospital
Locations (1):
- Geriatric Department, Broca Hospital, Paris, IIe-de-France, France